CLINICAL TRIAL: NCT06031740
Title: A Randomized Comparison of Flexible Endoscopic Polidocanol Liquid and Foam Sclerotherapy in Cirrhotic Patients With Bleeding From Internal Hemorrhoids
Brief Title: A Comparison of Flexible Endoscopic Polidocanol Liquid and Foam Sclerotherapy in Cirrhotic Patients With Bleeding From Internal Hemorrhoids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-63
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Liver Cirrhosis; Internal Hemorrhoid
MeSH Terms: conditions — Liver Cirrhosis | interventions — Sclerotherapy; Polidocanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sclerotherapy with 1.5% polidocanol. (Experimental): 2mL (3%) polidocanol = 60mg; maximal dose: 1mL/column and 4mL/session.
  Interventions: Procedure: Sclerotherapy with 1.5% polidocanol
- Foam sclerotherapy (Active Comparator): Tessari's technique; 4mL 3% poilidocanol +16mL air; maximal dose: 2mL/column and 20mL/session.
  Interventions: Procedure: Foam sclerotherapy.

INTERVENTIONS:
Procedure: Sclerotherapy with 1.5% polidocanol — 2mL (3%) polidocanol = 60mg; maximal dose: 1mL/column and 4mL/session.
  - Group 2: Foam sclerotherapy.
  Arms: Sclerotherapy with 1.5% polidocanol.
Procedure: Foam sclerotherapy. — Tessari's technique; 4mL 3% poilidocanol +16mL air; maximal dose: 2mL/column and 20mL/session.
  Arms: Foam sclerotherapy

SUMMARY:
Haemorrhoids are the most common proctologic disease, affecting up to 36% of people in the developed world. Sclerotherapy is deﬁned as the injection of sclerosing agents at the apex of the internal hemorrhoidal complex, above the dentate line, leading to scarring, ﬁbrosis, and ﬁxation of the hemorrhoids. Sclerotherapy as a treatment of internal hemorrhoids has been used for a long time by surgeons, using proctoscopic exposure. Even though flexible instruments can be expected to have better manoeuvrability and target site exposure. There is no consensus amongst the major guidelines as to which grade of haemorrhoid that sclerotherapy should be used, whether it is equivalent or inferior to rubber bad ligation (RBL), whether sclerotherapy should be used at all for the treatment of IH, what is the effect of PHT on hemorrhoid prevalence and propensity to bleed, differentiation of internal hemorrhoids from rectal varices, data on EBL or EST in cirrhotics with hemorrhoids, safety of endotherapy with underlying coagulopathy and concerns for infectious complications.

DETAILED DESCRIPTION:
Hypothesis :- Polidocanol foam sclerotherapy is more effective than liquid polidocanol sclerotherapy, for bleeding cessation from internal hemorrhoids in cirrhotic patients.

Aim and Objective - To compare flexible endoscopic polidocanol liquid and foam sclerotherapy in cirrhotic patients with bleeding from internal hemorrhoids

Primary objective: No recurrence of hemorrhoidal bleeding episodes at 1-week after endotherapy

Secondary objectives:

1. Ano-rectal bleeding at 4-wks, defined by Giamundo score. [Ordinal score 0-4]
2. Ano-rectal bleeding at 8-wks, defined by Giamundo score. [Ordinal score 0-4]
3. Proportion of patients requiring a 2nd treatment session within 8-wks. [Indications: Giamundo score >3, or hemoglobin drop >1g/dL, or requirement of transfusion, or clinician discretion; Time frame: 8-weeks]
4. Proportion of patients with failed endotherapy. [Persistent bleeding with Giamundo score >3 from internal hemorrhoids or treatment related ulcers, after 2nd endotherapy session; Time frame: 8-weeks]
5. Proportion of patients requiring BT for hemorrhoidal bleeding within 8 wks.
6. Relationship of MELD score (4-40) with no recurrence of bleeding at 7d.
7. Adverse events/ local infectious complications after endotherapy. [Time frame: 8-wks]
8. Proportion of cirrhotic patients with bleeding hemorrhoids, with coexisting rectal varices and/or portal colopathy.

Methodology:

- Study population: Patients with cirrhosis, attending outpatient clinics or admitted, with ano-rectal bleeding suspicious to be hemorrhoidal in origin. Investigator will include both compensated and decompensated (acute or chronic) cirrhotics with anorectal bleed, and patients with ACLF with ano rect1al bleed.

Study design: Open label, parallel group, randomized, controlled study.

* Study period: 1 year after IEC approval.
* Sample size with justification: Treatment success at 1-wk, after one liquid sclerotherapy session is expected in 50% cirrhotics.Treatment success after one session of foam sclerotherapy is expected in 85% cirrhotics. Assuming efficacy difference of 35%, significance (α) at 0.5, power of 80%, the two groups should include 27 patients each (Total 54). To compensate for dropouts, final sample size of 60 patients.
* Intervention:
* Cap-assisted, flexible endoscopic treatment in both groups.
* Group 1: Sclerotherapy with 1.5% polidocanol. 2mL (3%) polidocanol = 60mg; maximal dose: 1mL/column and 4mL/session.
* Group 2: Foam sclerotherapy. Tessari's technique; 4mL 3% poilidocanol +16mL air; maximal dose: 2mL/column and 20mL/session.
* Monitoring and assessment:
* Time of index procedure will be considered as baseline (T0). There will be three scheduled evaluation time points: At 1 week (T1), 4 weeks (T2), and at 8 weeks (T3).
* The degree of bleeding, prolapse, pain, quality of life, and patient satisfaction will be recorded at each visit.
* Statistical Analysis: The results will be reported as counts and percentages for categorical variables, and as mean ± SD (range) for continuous normally distributed variables and median (interquartile range [IQR]) for ordinal categorical variables and for continuous non-normally distributed variables. The chi-square test will be used for cross-tabulations. Continuous variables will be compared between the groups by using the Student's t test or the Mann-Whitney test, depending on the data distribution.The time to recurrence will be evaluated as the time elapsed from treatment success to the relapse of bleeding (at least 2 for the Giamundo bleeding score). Kaplan-Meier curves will be used to evaluate freedom from recurrence; statistical comparison of survival curves will be carried out by the log-rank test.The changes in the Giamundo score, and HDSS scores over time will be analyzed with the Friedman test, because these scores are not normally distributed. The results associated with a p-value <0.05 will be considered statistically significant.
* Adverse effects:
* The AEs will be classified as none, remote, possible, probable, or not assessable based on the relation with the sclerosant.
* Specific AEs to report:-

  1. Bleeding requiring Blood Tx, with hemodynamic instability or need for urgent surgery
  2. External thrombosis requiring surgical intervention
  3. Occurrence of urinary retention
  4. Prostatic infection
  5. Sexual dysfunction in men
  6. Perineal abscess
  7. Sepsis
* Stopping rule of study:
* Study will be stopped in case of life-threatening adverse event judged to be related to the protocol intervention at department review meeting.

  (c) Expected outcome of the project:
* Establishment of an effective treatment protocol for hemorrhoidal bleeding in cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhotic/ACLF patients with ano-rectal bleeding, either ongoing or within last 1-week, judged to be hemorrhoidal in origin based on clinical features and endoscopy evaluation.

Exclusion Criteria:

1. Coagulopathy threshold of INR >2.0 and/or platelet count <50,000/mm3.
2. Antiplatelet or anticoagulants use.
3. Immunosuppressive medications (including steroids >20mg/d or equivalent for >2 weeks).
4. Grade IV internal hemorrhoids.
5. Thrombosed or strangulated IH or EH.
6. Previous EST or RBL in last 1-year.
7. Co-existing ano-rectal diseases like perianal abscess, stricture, ﬁstula, anal malignancies, ano-rectal stenosis, radiation proctitis, or proctitis.
8. Patients not capable of understanding and signing the informed consent.
9. Pregnancy.
10. Bronchial Asthma.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-07 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with no recurrence of hemorrhoidal bleeding episodes at 1 week after endotherapy. | 1 week

SECONDARY OUTCOMES:
Number of participants with ano-rectal bleeding at 4 weeks, defined by giamundos core [ Ordinal score from 0-4 ; Higher score meaning worse outcome | 4 weeks
Number of participants with ano-rectal bleeding at 8 weeks, defined by giamundos core [ Ordinal score from 0-4 ; Higher score meaning worse outcome | 8 weeks
Proportion of patients requiring a 2nd treatment session within 8 weeks | 8 weeks
Proportion of patients with failed endotherapy. | 8 weeks
Proportion of patients requiring BT for hemorrhoidal bleeding within 8 weeks. | 8 weeks
Relationship of Model for end stage liver disease (MELD) score with no recurrence of bleeding at 7 days [ Minimum 4 to maximum 40; Higher meaning worse. | 7 days
Adverse events/ local infectious complications after endotherapy. | 8 weeks
Proportion of cirrhotic patients with bleeding hemorrhoids, with coexisting rectal varices and/or portal colopathy. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No